CLINICAL TRIAL: NCT04410887
Title: Neoadjuvant Chemotherapy With Pressurized Intra Peritoneal Aerosol Chemotherapy(PIPAC) Plus SOX Plus Olaparib (PISOXO) for Locally-invaded-gastric Cancer (LIGC)
Brief Title: Neoadjuvant Chemotherapy With PISOXO for Locally-invaded-gastric Cancer (LIGC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, BIRENDRA KUMAR SAH, Principal investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRAGON VI: PISOXO Phase I
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Stomach Cancer; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PISOXO (Experimental): 1. st cycle of PIPAC during 1st laparoscopic exploration Three cycles of SOX
  2. nd cycle of PIPAC during 2nd laparoscopic exploration Surgery Three cycles of SOX +/-OLAPARIB
  PIPAC Intraperitoneal chemotherapy for PIPAC is Docetaxel Neoadjuvant Chemotherapy Patients will receive three cycles of a standard dose of Tegafur gimeracil oteracil potassium capsule (TGO) plus oxaliplatin (SOX) +Olaparib prior to curative gastrectomy.
  Adjuvant chemotherapy Three cycles of SOX +/- OLAPARIB will be given as postoperative chemotherapy.
  Chemotherapy regimen A cycle consists of Day 1: Oxaliplatin 130mg/M2 intravenous Day 1-14 Tegafur gimeracil oteracil potassium capsule (TGO) 80mg/M2 oral (twice daily) Repeated every 21st day OLAPARIB Day 1-14: Olaparib 300mg oral twice a day
  Interventions: Drug: PIPAC+SOX+OLAPARIB

INTERVENTIONS:
Drug: PIPAC+SOX+OLAPARIB — SOX Chemotherapy regimen A cycle consists of Day 1: Oxaliplatin 130mg/M2 intravenous Day 1-14 Tegafur gimeracil oteracil potassium capsule 80mg/M2 oral (twice daily) Repeated every 21st day OLAPARIB Day 1-14: Olaparib 300mg BID PO
  Other Names: Chemotherapy

SUMMARY:
The main purpose of this study is to compare the safety and efficacy of PIPAC+SOX+OLAPARIB for locally-invaded-gastric cancer (LIGC) patients in China. To obtain preliminary results for designing a new phase II/III randomized controlled trial.

DETAILED DESCRIPTION:
Peritoneal metastases is the main cause of relapse and death after surgery in patients with serosa positive or locally-invaded-gastric cancer (LIGC). Recent researches showed that PIPAC and Olaparib are effective to control peritoneal metastases in different malignant diseases but it has not been tested for gastric cancer patients. The main purpose of this study is to compare the safety and efficacy of PIPAC+SOX+OLAPARIB for locally-invaded-gastric cancer (LIGC) patients in China. To obtain preliminary results for designing a new phase II/III randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Histology confirmed non-obstructive adenocarcinoma of the stomach or esophagogastric junction.
* Clinical stage: cTNM: T4b and or N0-3 M0
* Performance status: Eastern Cooperative Oncology Group (ECOG) ≤ 2 (normal to symptomatic but in bed less than half the day)
* Clinically fit for systemic chemotherapy and gastric cancer surgery, i.e. adequate renal, hepatic, hematologic, and pulmonary function.
* Written informed consent

Exclusion Criteria:

* Clinically unfit for systemic chemotherapy and gastric cancer surgery, i.e. uncontrolled cardiac disease, or other clinically significant uncontrolled comorbidities, unable to undergo general anesthesia
* Distant metastases
* Locally advanced inoperable disease (Clinical assessment)
* Relapse of gastric cancer
* Prior chemo or radiotherapy
* Inclusion in another clinical trial
* Known contraindications or hypersensitivity for planned chemotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | Upto three months after curative resection of the primary tumor
  Total percentage of patients with pathological complete or sub-total tumor regression (TRG1a+1b) in the primary tumour

SECONDARY OUTCOMES:
Overall survival (OS) | Five years
  Overall survival (OS): Time from randomization to death from relapse
Disease free survival (DFS) | Three years
  Time from randomization to relapse of disease

CONTACTS AND LOCATIONS:
Overall Officials: Birendra K Sah, PH D, Principal Investigator — Ruijin Hospital; Chen Li, PH D, Study Director — Ruijin Hospital; Zhenggang Zhu, PH D, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No